CLINICAL TRIAL: NCT00130650
Title: Efficacy of Pain Ease Spray in Reducing Needle Pain Associated With Intravenous Insertion in Children
Brief Title: Pain Ease Spray in Reducing Needle Pain Associated With Intravenous Insertion in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: William Splinter, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05/31E
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Pain
Keywords: IV; cannulation; Injections, Intravenous
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pain Ease

SUMMARY:
The purpose of this study is to investigate the use of a new vapocoolant spray, Pain Ease, to reduce intravenous (IV) insertion pain in school-aged children receiving treatment in the Emergency Department.

DETAILED DESCRIPTION:
Inserting a needle into a child's vein is a distressing experience for children. Reducing the pain of injection and avoiding the child's discomfort remains an important aim for both parents and health care workers. Withdrawing blood and intravenous insertion (IV) in children is also time consuming, especially when the child is uncooperative and stressed.

We, the researchers at Children's Hospital of Eastern Ontario, have been searching for an effective, rapid and inexpensive method to alleviate the distress associated with venipuncture and IV insertion.

Medications by mouth, such as anti-anxiety drugs, are helpful but usually do not significantly reduce the pain. The most commonly used anti-anxiety drug at our institution is midazolam, but unfortunately onset of action takes 20-30 minutes. There are various forms of topical creams that can numb the skin. EMLA, a mixture of two local anesthetics (Lidocaine 2.5% and Prilocaine 2.5%), is applied as a topical cream and is covered with an occlusive dressing. It requires at least 1 hour to be effective. It is not only time consuming but expensive (~$1.30 per application). Ametop (Tetracaine PH. Eur.4%w/w) is another effective topical cream, which works in 30 minutes, but it is more expensive than EMLA (~$3.00 per application). Vapocoolant sprays applied for ~10 seconds immediately before injection have been shown to be faster, less expensive and as effective as EMLA in reducing pain at the site of injection during immunization.

The current investigation will evaluate the quality, efficacy and costs associated with the use of a new vapocoolant spray, Pain Ease, in reducing pain associated with IV insertion for school age children.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* Require an IV inserted in less than 30 minutes

Exclusion Criteria:

* Allergy to vapocoolant sprays
* Vascular impairment
* Diabetes mellitus
* Developmental delay/inability to understand pain scale
* Received analgesia in last 24 hours
* Triaged as resuscitation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
pain score | at injection (< 1 minute)

SECONDARY OUTCOMES:
anxiety score | at injectiong (< 1 minute)
satisfaction (nurse, parent) | <10 minutes post-injection
IV insertion time | immediate
ease of IV insertion | immediate

CONTACTS AND LOCATIONS:
Overall Officials: William M Splinter, BSc, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Farion KJ, Splinter KL, Newhook K, Gaboury I, Splinter WM. The effect of vapocoolant spray on pain due to intravenous cannulation in children: a randomized controlled trial. CMAJ. 2008 Jul 1;179(1):31-6. doi: 10.1503/cmaj.070874. PMID 18591524